CLINICAL TRIAL: NCT07156331
Title: Research on Effects of Drugs on Body Composition and Function With Imaging in Diabetes
Acronym: REBUILD
Status: Not yet recruiting | Type: Observational
Sponsor: Kristin Clemens (Other)
Responsible Party: Sponsor-Investigator, Kristin Clemens, Associate Professor, Western University, Canada
Organization: Western University, Canada (Other)
Other Study IDs: REBUILD
Record Dates: First submitted 2025-08-07; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: T2DM; Type 2 Diabetes; Semaglutide; Tirzepatide; GLP-1RA; GLP-1RA/GIP; Body Mass; Muscle Composition; Muscle Mass; Mounjaro; Ozempic; Wegovy; DM2; Diabetes Mellitus 2; Muscle Strength; Muscle Function; Muscle Preservation; Bone Health
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with T2DM that have recently been started on GLP-1RA or GLP-1RA/GIP Medication: Adults at least 18 years of age that have Type 2 Diabetes, have recently been started on semaglutide or tirzepatide under the care of a physician

SUMMARY:
One downside of diabetes weight loss drugs like GLP-1RA and GLP-1RA/GIP, is that they can cause muscle loss, which is especially risky for older adults or those already prone to frailty and falls. There is also concern that GLP-1RA might affect bone health, possibly leading to weaker bones and increased risk of fractures. To prevent these issues, doctors need to better predict who is most at risk of muscle and/or bone loss. That way, doctors can adjust patient management-like adding targeted physical therapy, or bone-protecting medications alongside GLP-1RA or GLP-1RA/GIP medications.

Medical imaging can help spot early muscle and bone changes. Advanced imaging, like PET and CT scans allow for the assessment of muscle fat content and blood flow in the bones and muscles. This could provide clearer insights into how GLP-1RA or GLP-1RA/GIP medications affect muscles and bones in ways that matter for patients (strength, mobility, falls risk, etc.).

The investigators will conduct an exploratory study of 20 patients initiating on GLP-1RA or GLP-1RA/GIP by their care provider, and assess their muscle and bone health at baseline, 3, 6, and 12 months using advanced PET/CT imaging. The investigators will also assess functional measures, including grip strength, Timed Up and Go test, and gait speed. The goal is to measure and describe early changes in body composition and physical function that could signal harm. These findings will help to develop a clinical prediction tool for clinicians to use prior to starting semaglutide or tirzepatide, as well as design interventions to help promote healthy muscle and bone while on treatment.

DETAILED DESCRIPTION:
In Canada, older adults are projected to represent nearly one-fourth of the population by 2040, with the number of old older adults (75 and older) growing at an even faster rate. This demographic shift has important implications, including a rising prevalence of aging-related disease. Approximately 1 in 4 Canadians aged 65 or older have type 2 diabetes (DM2).

Aging and DM2 often coexists with obesity, chronic kidney disease (CKD) and/or cardiovascular disease (CVD) as well as cardiovascular-kidney-metabolic (CKM) syndrome. Aging and chronic disease also independently elevate the risk of sarcopenia (age-related progressive loss of muscle mass and strength) and frailty.

Glucagon-like peptide 1 receptor agonists (GLP-1RA like Ozempic) have revolutionized the management of chronic metabolic disease. These agents lower blood glucose, promote weight loss, and protect the heart, brain, and kidneys, making them the cornerstone of therapy for diabetes, kidney, cardiovascular, and CKM syndrome. However, concerns have been raised about the amount of weight loss elicited by these medications, particularly the associated loss of skeletal muscle mass. In some studies, weight loss of greater than 10 kg have been described with GLP-1RA (i.e., semaglutide) or GLP-1RA/GIP (tirzepatide) drugs, with up to 40% of total weight loss from lean body mass reported with semaglutide. Loss of lean body mass (including skeletal muscle mass), could be particularly worrisome to those at high risk for frailty and sarcopenia, both of which are associated with increased morbidity, hospitalizations, reduced quality of life, disability and mortality. There is also evidence that these medications could negatively impact bone quality and fracture risk.

Existing studies on the impact of GLP-1RA and GLP-1RA/GIP on lean body mass have been limited; they primarily measured body composition using dual energy x ray absorptiometry (DXA) which is unable to quantify intramuscular fat, and is less sensitive to body thickness and hydration/pathologic status. DXA also has lower precision/accuracy compared with CT scan and MRI, leading to more variability. Among studies that have used MRI to examine body composition, many were secondary analyses of clinical trials, excluded individuals with body mass index (BMI) ≤25 kg/m2 and/or DM2, had short follow-up, and lacked functional assessments. Evidence indicates that intramuscular fat is more strongly associated with adverse outcomes than muscle quantity, highlighting the importance of exploring the impact of GLP-1RA and GLP-1RA/GIP on both muscle mass and muscle composition. There also remains an opportunity to examine the association between changes in body composition and measures of muscle strength/function, which are highly prognostic of outcomes such as disability, hospitalizations, and mortality. There is also a dearth of evidence regarding the impact of GLP-1RA and GLP-1RA/GIP medications on muscle blood flow, glucose metabolism, or bone blood flow, which may correlate with clinically important patient outcomes like falls and fracture.

The investigators propose a single-arm, open-label, prospective study to explore changes in body composition, muscle mass, composition, and function, in patients with DM2 with and without CKM following initiation of a GLP-1RA (semaglutide or Ozempic is the most commonly prescribed) or GLP-1RA/GIP (tirzepatide or Mounjaro is the most commonly prescribed). The goal is to characterize and quantify early changes in muscle and physical function that could signal harm; This will allow the development clinical prediction tool to guide treatment decisions before initiating semaglutide or tirzepatide, and to design targeted interventions aimed at preserving muscle and bone health in real-world patients with type 2 diabetes prescribed GLP-1RA or GLP-1RA/GIP therapies.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have type 2 diabetes
* Have recently been started on semaglutide or tirzapatide under the care of a physician
* Be able to speak and read English

Exclusion Criteria:

* Are pregnant or breastfeeding
* Are unable to perform functional tests
* Are unable to provide informed consent
* Have any contraindication to PET/CT scan
* Had a change in body weight over 5 kilograms within 90 days before starting a GLP-1RA or GLP-1RA/GIP
* Had previous or planned (during the study period) bariatric surgery in the subsequent 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 or older with type 2 diabetes that have recently been started on semaglutide or tirzepatide under the care of a physician.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle mass at 1-year | Change from baseline to 12 months
  Changes in skeletal muscle mass 1-year after initiation semaglutide or tirzepatide. Measured at the L3 lumbar vertebrae with PET-CT, in cm²/m².
Change in Timed Up-and-Go (TUG) at 1-year | Change from baseline to 12 months
  Change in muscle strength and function 1-year after starting semaglutide or tirzepatide. Measures the time in seconds to stand from a standard chair, walk 3 meters, turn, walk back and sit down. Measured in seconds.
Change in Gait Speed at 1-year | Change from baseline to 12 months
  Change in muscle strength and function 1-year after starting semaglutide or tirzepatide. Usual-pace walking speed measured across a 4-meter course with a static start. Measured in meters per second.
Change in Handgrip Strength at 1-year | Change from baseline to 12 months
  Change in muscle strength - handgrip strength change 1-year after starting semaglutide or tizepatide. Measured using handheld dynamometer in the dominant hand, in kg.

SECONDARY OUTCOMES:
Change in skeletal muscle quality at 3 and 6 months | Change from baseline to 3 months, change from baseline to 6 months
  Changes L3 skeletal muscle radiodensity 3 months and 6 months after initiation of semaglutide or tirzepatide. Measured at L3 lumbar vertebrae with PET-CT, in Hounsfield Units (HU).
Change in skeletal muscle quality at 3 and 6 months | Change from baseline to 3 months, change from baseline to 6 months
  Changes L3 skeletal muscle radiodensity at 3 months and 6 months after initiation of semaglutide or tirzepatide. Measured at L3 lumbar vertebrae with PET-CT, in Hounsfield Units (HU).
Change in Timed Up-and-Go (TUG) at 3 and 6 months | Change from baseline to 3 months, change from baseline to 6 months
  Change in muscle strength and function 3 months and 6 months after starting semaglutide or tirzepatide. Measures the time in seconds to stand from a standard chair, walk 3 meters, turn, walk back and sit down. Measured in seconds.
Change in Gait Speed at 3 and 6 months | Change from baseline to 3 months, change from baseline to 6 months
  Change in muscle strength and function 3 months and 6 months after starting semaglutide or tirzepatide. Usual-pace walking speed measured across a 4-meter course with a static start. Measured in meters per second.
Change in Handgrip Strength at 3 and 6 months | Change from baseline to 3 months, change from baseline to 6 months
  Change in muscle strength - handgrip strength change 3 months and 6 months after starting semaglutide or tizepatide. Measured using handheld dynamometer in the dominant hand, in kg.

OTHER OUTCOMES:
Blood Flow in Muscle, Bone and Kidney | 12 months
  Changes in blood flow in muscle, bone and kidney 1 year after starting semaglutide or tirzepatide.
Glucose Metabolism in Muscle, Bone and Kidney | 12 months
  Changes in glucose metabolism in muscle, bone and kidney 1 year after initiating semaglutide or tirzepatide.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Clemens, MD, MSc, Principal Investigator — St. Joseph's Health Care London

IPD SHARING:
Plan to Share IPD: No